CLINICAL TRIAL: NCT01893736
Title: A Randomized Controlled Trial of a Professional Breastfeeding Support Intervention to Increase the Exclusivity and Duration of Breastfeeding
Brief Title: Professional Breastfeeding Support Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Marie Tarrant, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBFS-1
Record Dates: First submitted 2013-06-06; First posted 2013-07-09 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Breastfeeding
Keywords: Breastfeeding; professional support; postnatal; interventions; exclusive breastfeeding; randomized controlled trial
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): In-hospital usual care consists of routine intrapartum and postnatal obstetric care. No extra intervention will be provided by research team.
- In-hospital professional support (Experimental): The participants in "in-hospital professional support" arm will receive three 30-minute one-to-one hands-on breastfeeding counseling sessions during postpartum hospitalization.
  Interventions: Other: In-hospital professional support
- Postpartum telephone follow-up support (Experimental): Participants in "postpartum telephone follow-up support" arm will receive telephone support in the first 4 weeks postpartum.
  Interventions: Other: Postpartum telephone follow-up support

INTERVENTIONS:
Other: In-hospital professional support — In-hospital professional lactation support will consist of two 30-minute one-to-one hands-on breastfeeding counseling sessions in first 24 hours post-partum and one further 30-minute one-to-one hands-on breastfeeding counseling session on the second day of post-partum hospitalization for a total of three 30-minute sessions. The one-to-one sessions will focus on: (1) education and advice on correct breastfeeding positions and techniques, (2) education and advice on milk supply and how to avoid common breastfeeding problems, and (3) hands-on instruction and assistance with proper breastfeeding positioning and technique, latching on and newborn attachment to the breast, and manual expression of breast milk.
  Arms: In-hospital professional support
Other: Postpartum telephone follow-up support — Postpartum telephone follow-up support will consist of telephone support 72 hours after hospital discharge and weekly for the first 4 weeks, or until weaned. Earlier telephone contacts will focus more on breastfeeding topics. Information will be solicited from the participants about problems or difficulties they are experiencing. Supportive advice will be provided regarding management of breastfeeding problems, and support and encouragement for the continuation of breastfeeding. Later contacts will focus more on advice and encouragement on breastfeeding while resuming daily activities or returning to work, nursing in public places, and expressing and storing breast milk.
  Arms: Postpartum telephone follow-up support

SUMMARY:
The investigators will conduct an early postpartum professional breastfeeding intervention to postpartum women who are intended to breastfeed newborn babies to improve breastfeeding outcomes.

DETAILED DESCRIPTION:
The aim of this study is to determine whether early post-partum professional breastfeeding support improves breastfeeding outcomes.

The primary hypotheses are:

1. Exclusive breastfeeding rates at 1, 2, and 3 months will be increased among mother-infant pairs who receive professional lactation support or telephone follow-up support (intervention groups) when compared with those who receive usual post-natal breastfeeding support (control group);
2. The rate of any breastfeeding (predominant or partial) at 1, 2, and 3 months will be increased among mother-infant pairs in the intervention groups when compared with those in the control group;

The secondary hypotheses are:

1. The overall duration of exclusive breastfeeding will be increased among mother-infant pairs in the intervention groups when compared with those in the control group;
2. The overall duration of any breastfeeding (predominant or partial) will be increased among mother-infant pairs in the intervention groups when compared with those in the control group.

ELIGIBILITY:
Inclusion Criteria:

1. delivers at participating trial site,
2. primiparous,
3. intends to breastfeed,
4. 18 years of age or older,
5. has singleton pregnancy,
6. Cantonese speaking,
7. Hong Kong resident for more than one year,
8. no serious medical or obstetrical complications

Exclusion Criteria:

1. < 37 weeks gestation,
2. an Apgar score < 8 at five minutes,
3. a birth weight < 2500 grams,
4. born with any severe medical conditions or congenital malformations,
5. is placed in the special care nursery for more than 48 hours after delivery,
6. is placed in the intensive care nursery after delivery,
7. not entitled to health benefits in Hong Kong (NEP).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of any and exclusive breastfeeding | 1 month postpartum
  Any breastfeeding rate and exclusive breastfeeding rate at 1 month postpartum
Prevalence of any and exclusive breastfeeding | 2 months postpartum
  Any breastfeeding rate and exclusive breastfeeding rate at 2 months postpartum
Prevalence of any and exclusive breastfeeding | 3 months postpartum
  Any breastfeeding rate and exclusive breastfeeding rate at 3 months postpartum

SECONDARY OUTCOMES:
Median duration of breastfeeding | 6 month postpartum
  The median duration of any breastfeeding and the median duration of exclusive breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Tarrant, PhD, MPH, RN, Principal Investigator — The University of Hong Kong
Locations (4):
- Hong Kong (4):
  - Kwong Wah Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong

REFERENCES:
- [Result] Fu IC, Fong DY, Heys M, Lee IL, Sham A, Tarrant M. Professional breastfeeding support for first-time mothers: a multicentre cluster randomised controlled trial. BJOG. 2014 Dec;121(13):1673-83. doi: 10.1111/1471-0528.12884. Epub 2014 May 26. PMID 24861802